CLINICAL TRIAL: NCT05148130
Title: Construction and Biological Study of Blood and Placenta Samples Associated With Gestational Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-121
Record Dates: First submitted 2021-06-27; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-06

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — maternal peripheral blood; blood serum after centrifugation; DNA extracted from the peripheral blood; umbilical cord blood; the placenta tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the gestational diabetes pregnant women group: The diagnosis of GDM was established following the International Association of Diabetes and Pregnancy Study Groups (IADPSG) diagnostic criteria. GDM should be diagnosed at any time in pregnancy if one or more of the listed criteria are met following a 75-gram glucose load: fasting plasma glucose ≥5.1 mmol/l, 1-hour plasma glucose ≥10.0 mmol/l, and 2-hour plasma glucose of 8.5-11.0 mmol/l. Women diagnosed with DM or prediabetes (impaired fasting glucose or impaired glucose tolerance) before pregnancy were excluded from the study.
  Interventions: Diagnostic Test: oral glucose tolerance test
- the healthy pregnant control group: the control group was pregnant women who delivered a single fetus at full term without complications and complications during pregnancy
  Interventions: Diagnostic Test: oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: oral glucose tolerance test — GDM should be diagnosed at any time in pregnancy if one or more of the listed criteria are met following a 75-gram glucose load: fasting plasma glucose ≥5.1 mmol/l; 1-hour plasma glucose ≥10.0mmol/l; 2-hour plasma glucose 8.5-11.0 mmol/l. Those women diagnosed with diabetes or pre-diabetes (impaired fasting glucose or impaired glucose tolerance) before pregnancy were excluded from the study.

SUMMARY:
Gestational diabetes mellitus (GDM) is a type of diabetes mellitus with normal glucose metabolism before pregnancy. Pregnant women with prepubertal diabetes have complicated clinical experiences, and the effects of severe disease or poor glycemic control on mothers and infants. The incidence of gestational diabetes mellitus is very high, and the short-term and long-term complications of the mother and the child are higher. Through the detection of blood samples, we can not only obtain the basic information related to the disease such as blood cells and blood biochemistry, but also learn the important information such as enzymes, antibodies and cell metabolites in the blood that are conducive to the diagnosis of the disease. More importantly, blood contains genetic material (such as genomic DNA) that can be used to screen for genes and break down molecules. Placenta tissue examination can provide important cellular, biochemical, immunological and other information. However, due to the complex etiology of gestational diabetes. Especially associated with genetic or immunological factors, in the short term often cannot make a definite diagnosis, and patients in hospital time is limited, some check items such as gene detection, placental tissue can't complete them in hospital, need to return the patient's blood, cord blood and placenta tissue, to facilitate later further screening and biology research. This study intended to establish gestational diabetes patient's blood, cord blood and placenta tissue samples library, screening is closely related to the disease biomarkers, such as disease-causing gene mutations, susceptible gene mutation and protein metabolism product, so as to clarify disease relationship between genotype and clinical phenotype, the pathogenesis of diseases, etc., and provide the basis for the diagnosis of disease and treatment optimization.

DETAILED DESCRIPTION:
the registry procedures: we collected data and blood samples from pregnant women diagnosed with GDM and matched healthy pregnant women as controls on the day admitted to hospital for delivery. All of the participants recruited were Han Chinese. Placental tissue was collected immediately after delivery and saved at -20 °C for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient was older than 18 years old and had not been diagnosed with diabetes before pregnancy. A 75-gram glucose load examination was performed during 24-28 weeks of gestation：GDM should be diagnosed at any time in pregnancy if one or more of the listed criteria are met following a 75-gram glucose load: fasting PG ≥5.1 mmol/l; 1-hour PG ≥10.0mmol/l; 2-hour PG 8.5-11.0 mmol/l.
2. If the patient is younger than 18 years old, consent from parents or guardians is required;
3. Inclusion objects in line with the above sample sources;
4. Signed the informed consent;

Exclusion Criteria:

1. Refuse to sign the informed consent
2. Severe mental symptoms, unable to cooperate with blood collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All of the subjects come from the Department of Obstetrics of Second Hospital Affiliateod to Zhejiang University Medical College, Hangzhou, Zhejiang Province。
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2022-09-11 (Estimated); Study Completion 2023-09-11 (Estimated)

PRIMARY OUTCOMES:
glucose homeostasis levels | 1 year
  fasting plasma glucose, 1-hour plasma glucose and 2-hour plasma glucose in mmol/l
genotype of GDM single gene polymorphism | 1 year
  genotype such as the Surfactant protein-D gene polymorphism rs721917 in Thr31Met
blood biochemistry indices | 1 year
  such as the serum Surfactant protein-D protein levels in ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Li Q Wang, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Zhenjiang, China

IPD SHARING:
Plan to Share IPD: Undecided
At present, we only share partial data of patients with gestational diabetes: blood glucose, BMI, age, fetal birth weight and other general features。